CLINICAL TRIAL: NCT01582750
Title: Endoscopic Ultrasound Predict the Sensitivity of Stage II / III Rectal Cancer Preoperative Concurrent Chemoradiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., Director of Abdomen Division, Radiation Oncology Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CH-RO-GI-eus
Record Dates: First submitted 2012-04-19; First posted 2012-04-23 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Rectal Cancer
Keywords: endoscopic ultrasound; pre-operative concurrent chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Local advanced rectal cancer EUS

SUMMARY:
The purpose of this study is to determine the role of endoscopic ultrasound measurement of the primary tumor maximum diameter changes in absolute / relative values in predicting the tumor regression after concurrent chemoradiotherapy for rectal cancer.

DETAILED DESCRIPTION:
We use endoscopic ultrasound to measure the primary tumor maximum diameter changes to predict the tumor regression after concurrent chemoradiotherapy for rectal cancer

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed rectal cancer, preoperative stage II / III (T3-4N0 or T1-4N + M0).
* tumor distance from anus less than 12 cm.
* KPS score not less than 70
* can be tolerated chemotherapy and radiotherapy.
* pelvic who had no history of radiation therapy.
* Non-allergic history of fluorouracil or platinum-based chemotherapy drugs.
* a full understanding of the study, the ability to complete all of the treatment plan, follow up the conditions and sign the informed consent.

Exclusion Criteria:

* other malignancy (past or at the same time), does not include curable non-melanoma skin cancer and cervical carcinoma in situ; does not include resectable primary colon cancer (synchronous or metachronous).
* pregnant or lactating patients.
* fertility but did not use contraceptive measures.
* existing active infection.
* merge serious complications, can not tolerate the treatment, such as 6 months of myocardial infarction, mental illness, uncontrollable diabetes or uncontrollable hypertension or hypotension.
* concurrent treatment with other anticancer drugs.
* can not complete treatment or follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local advanced rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Endoscopic ultrasound measurement of the primary tumor maximum diameter changes in absolute / relative values | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, M.D., Principal Investigator — Chinese Acedemy of Medical Sciences
Locations (1):
- Li Ning, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li N, Dou L, Zhang Y, Jin J, Wang G, Xiao Q, Li Y, Wang X, Ren H, Fang H, Wang W, Wang S, Liu Y, Song Y. Use of sequential endorectal US to predict the tumor response of preoperative chemoradiotherapy in rectal cancer. Gastrointest Endosc. 2017 Mar;85(3):669-674. doi: 10.1016/j.gie.2016.06.042. Epub 2016 Jun 25. PMID 27354104